CLINICAL TRIAL: NCT00005892
Title: Study of Allogeneic Bone Marrow Transplantation Following Cyclophosphamide and Radiotherapy in Patients With Myelodysplastic Syndrome and Acute Leukemia Related to Fanconi's Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fairview University Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15100; UMN-MT-1985-01; UMN-MT-8501
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Fanconi's Anemia; Myelodysplastic Syndromes; Leukemia, Nonlymphocytic, Acute; Leukemia, Lymphocytic, Acute
Keywords: Fanconi's anemia; acute leukemia; acute lymphocytic leukemia; acute myeloid leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia; adult acute myeloid leukemia in remission; aplastic anemia; childhood acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia; childhood acute myeloid leukemia in remission; de novo myelodysplastic syndrome; hematologic disorders; hematopoietic/lymphoid cancer; leukemia; myelodysplastic syndrome; oncologic disorders; previously treated myelodysplastic syndrome; rare disease; secondary myelodysplastic syndrome
MeSH Terms: conditions — Fanconi Anemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Anemia, Aplastic; Hematologic Diseases; Hematologic Neoplasms; Leukemia; Rare Diseases | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide
Procedure: Allogeneic Bone Marrow Transplantation

SUMMARY:
OBJECTIVES:

I. Determine the effectiveness of moderate dose cyclophosphamide and radiotherapy in terms of improving survival and reducing the morbidity following allogeneic bone marrow transplantation in patients with myelodysplastic syndrome and acute leukemia related to Fanconi's anemia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive cyclophosphamide IV over 1-2 hours on day -6 through -3 and total body radiotherapy on day -1. Patients undergo allogeneic bone marrow transplantation on day 0.

ELIGIBILITY:
* Diagnosis of Fanconi's anemia with the family history and typical phenotype including: Short stature Hypoplastic radii Skin pigmentation Renal anomalies Chromosomal fragility
* Evidence of Fanconi's myelodysplastic syndrome Bone marrow dysplasia of all 3 marrow cell lines AND Clonal cytogenetic abnormalities demonstrable in marrow cells
* First complete remission following therapy for Fanconi's acute leukemia allowed
* Must have related histocompatible donor No evidence of excessive in vitro chromosome fragility typical of Fanconi's anemia Normal CBC and bone marrow

Ages: 0 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, Study Chair — Fairview University Medical Center
Locations (1):
- Fairview University Medical Center, Minneapolis, Minnesota, United States